CLINICAL TRIAL: NCT06879249
Title: The Effect of Critical Ultrasonography Guided Precise Fluid Management in Patients With Sepsis or Septic Shock: A Single-center Randomized Controlled Trial
Brief Title: The Effect of CUGP Fluid Management in Patients With Sepsis or Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shusheng Li (Other)
Responsible Party: Sponsor-Investigator, Shusheng Li, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEPSIS-CUGP; YLGX-ZZ-2020001 (Other Grant/Funding Number: The China Primary Health Care Foundation)
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-03

CONDITIONS: Sepsis
Keywords: sepsis, septic shock, fluid management, critical ultrasonography, volume responsiveness
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CUGP group (Experimental): In the CUGP group, ultrasonographic assessment was performed by a team of trained critical ultrasonography physicians at enrollment, 1 hour, 3 hours, 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours thereafter, respectively.
  Interventions: Device: critical ultrasonography
- usual care group (No Intervention): The usual care group used conventional hemodynamic monitoring methods for monitoring and decision-making about fluid management. Records were made at enrollment, 1 hour, 3 hours, 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours thereafter, respectively.

INTERVENTIONS:
Device: critical ultrasonography — In the CUGP group, attending physicians utilized a designed fluid management strategy guided by ultrasonographic evaluation of the inner diameter of IVC, ejection fraction (EF) value and passive leg raising-induced changes in VTI (ΔVTI). This ultrasonographic assessment was performed by a team of trained critical ultrasonography physicians at enrollment, 1 hour, 3 hours, 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours thereafter, respectively. Additionally, patients did not preclude the concurrent use of conventional hemodynamic monitoring methods. At each of these time points, attending physicians would make comprehensive decisions on fluid management based on the results of ultrasonographic evaluation, along with other monitoring methods. The researcher recorded the basis of decisions, disposal strategy and outcomes.
  Arms: CUGP group

SUMMARY:
This study aims to assess whether procedural critical ultrasonography guided precise fluid management (CUGP) can affect the clinical fluid management strategy and improve the outcomes of patients with sepsis or septic shock.

DETAILED DESCRIPTION:
This single-center parallel randomized controlled trial aims to assess whether procedural critical ultrasonography guided precise fluid management (CUGP) can affect the clinical fluid management strategy and improve the outcomes of patients with sepsis or septic shock. We planned to conduct this single-center trial in the intensive care unit (ICU) of Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology in Wuhan, China. Patients, who are initially diagnosed with sepsis, will be assessed for eligibility immediately upon admission to the ICU. Then, eligible participants will be informed and randomly assigned to one of the two groups: the CUGP group or the usual care group, in a 1:1 ratio using block randomization. In the CUGP group, ultrasonographic assessment was performed by a team of trained critical ultrasonography physicians at enrollment, 1 hour, 3 hours, 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours thereafter, respectively. The usual care group used conventional hemodynamic monitoring methods for monitoring and decision-making about fluid management. The enrolled patients received either CUGP or usual care fluid management within 72 hours of enrollment in the ICU, and followed by 60 days after randomization. The primary outcome was the 60-day all-cause mortality. The secondary outcomes included SOFA score at 24, 48, and, 72 hours after enrollment, fluid infusion volume, vasoactive drug dosage, incidence of serious adverse events related to fluid management, including new tracheal intubation, severe acute kidney injury, electrolyte disturbance, and organ ischemia (brain, myocardium, gastrointestinal tract, limbs), incidence of complications related to central venous and arterial puncture, acute left heart failure, and pulmonary edema, monitoring failure rates of CUGP group and usual care group, ICU and hospital length of stay, cost of ICU stay/hospitalization. This study adopts a standardized data collection and management system. The study implementer shall fill in the paper or electronic CRF.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old;
* 2. Estimated length of ICU stay ≥ 24 hours;
* 3. Diagnosis according to the Sepsis 3.0 criteria, which included:
* a. suspected or confirmed infections supported by clinical evidence and/or positive microbiological findings;
* b. the sepsis related organ failure assessment (SOFA) score ≥ 2.

Exclusion Criteria:

* 1. Patients were pregnant woman;
* 2. Patients had acute coronary syndrome;
* 3. Patients had acute pulmonary edema;
* 4. Patients had status asthmatics;
* 5. Patients had malignant arrhythmia;
* 6. Patients had active gastrointestinal bleeding;
* 7. Patients had epileptic seizure;
* 8. Patients had drug poisoning;
* 9. Patients had severe burns;
* 10. Patients had contraindications of blood transfusion;
* 11. Patients had intra-abdominal hypertension (intra-abdominal pressure increases continuously ≥ 12mmHg);
* 12. Patients had acute pulmonary embolism;
* 13. Patients had contraindications of leg raising;
* 14. Patients had cardiac structural or functional abnormalities (left ventricular outflow tract obstruction, moderate-to-severe mitral regurgitation, aortic regurgitation), it would seriously affect the velocity time integral of left ventricular outflow tract;
* 15. Patients or their legal representatives refused active treatment;
* 16. Patients or their legal representatives refused to participate in this study;
* 17. Patients were participating in other interventional clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-01-28 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
60-day all-cause mortality | At day 60 after randomization
  It refers to the total number of patients who died from any cause within 60 days of enrollment. It will be described as a rate

SECONDARY OUTCOMES:
72-hour SOFA Score | At baseline (before randomization), 24 hours, 48 hours, and 72 hours thereafter.
  The SOFA (Sequential Organ Failure Assessment) score was based on six different scores, one for each of the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems each scored from 0 to 4 with an increasing score reflecting worsening organ dysfunction.
Fluid management for decision | Within 72 hours of admission
  It included monitoring failure rates in the CUGP and usual care groups. In the CUGP group, monitoring failure was recorded if ultrasonographic results conflicted with conventional hemodynamic monitoring or if fluid management based on ultrasonography led to severe complications due to volume inadequacy or overload. Failure was also noted if management based on conventional monitoring improved hemodynamics. Additionally, inability to perform ultrasonography due to factors such as obesity, subcutaneous emphysema, or poor image quality was classified as failure. Patients with monitoring failure and severe complications were promptly transferred to the usual care group for safety. In the usual care group, monitoring failure was recorded if patients could not undergo conventional monitoring or if severe complications occurred following fluid management based on conventional methods. These patients were promptly transferred to the CUGP group to reduce risks.
Complications | Within 72 hours of admission
  It includes the incidence of complications related to central venous and arterial puncture, nosocomial infection, acute left heart failure, pulmonary edema, etc..
Fluid changes with 72 hours | Within 72 hours of admission
  Record the changes in fluid within 72 hours after admission
Dosage of vasopressors changes with 72 hours | Within 72 hours of admission
  Record the changes in dosage of vasopressors within 72 hours after admission
Survival time | Follow-up after 60th day after enrollment
  The survival time of patients was followed up 60th day after enrollment.
Length of ICU stays/hospitalization | Follow-up 60th day after enrollment
  The length of ICU stays/hospitalization patients was followed up 60th day after enrollment.
Cost of ICU stays/hospitalization | Follow-up 60th day after enrollment
  The cost of ICU stays/hospitalization patients was followed up 60th day after enrollment.
Serious adverse events | Follow-up 60th day after enrollment
  Serious adverse events occurred after enrollment. Tracheal intubation was defined as new intubation, and non-invasive mechanical ventilation as new usage after enrollment. Severe acute kidney injury was defined as a creatinine increase to three times the baseline or above 354 µmol/L, or the initiation of renal replacement therapy (RRT), excluding patients with chronic kidney failure on long-term dialysis. RRT referred to new use in patients without a history of long-term dialysis. Hypernatremia was defined as serum sodium above 159 mmol/L, and hyperchloremia as serum chloride above 115 mmol/L. Cerebral ischemia/infarction was identified by CT or MRI, while myocardial ischemia/infarction was defined by acute coronary syndrome, ischemic signs on ECG, or the need for coronary intervention or antithrombotic therapy. Intestinal ischemia was confirmed by endoscopy, surgery, or CT angiography, and limb ischemia was indicated by severe mottling and ischemia in the limbs.
Nosocomial infection during ICU stays | Follow-up 60th day after enrollment
  The Nosocomial infection during ICU stays was followed up 60th day after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Shusheng Li, PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Critical Care Medicine, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
IPD after de-identification can be shared on individual request to the principal investigator at lishusheng@hust.edu.cn.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available for two years after the publication of the primary outcomes.